CLINICAL TRIAL: NCT06993922
Title: Dexmedetomidine as an Adjuvant to Bupivacaine in Scalp Block Versus Bupivacaine Alone for Postoperative Pain Management in Patients Undergoing Craniotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Omar Ahmed Zakaria Khiralla, Resident of Anaesthesia, Intensive Care Unit and Pain, Faculty of Medicine, Ain shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MS 57/2025
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Dexmedetomidine; Adjuvant; Bupivacaine; Scalp Block; Postoperative Pain; Craniotomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group SB (Active Comparator): Patients will receive a scalp block with bupivacaine alone.
  Interventions: Other: Scalp block
- Group SD (Experimental): Patients will receive a scalp block with dexmedetomidine as an adjuvant to bupivacaine.
  Interventions: Other: Scalp block + Dexmedetomidine

INTERVENTIONS:
Other: Scalp block — Patients will receive a scalp block with bupivacaine alone.
  Other Names: Bupivacaine
  Arms: Group SB
Other: Scalp block + Dexmedetomidine — Patients will receive a scalp block with dexmedetomidine as an adjuvant to bupivacaine.
  Other Names: Bupivacaine + Dexmedetomidine
  Arms: Group SD

SUMMARY:
This study aims to compare dexmedetomidine as an adjuvant to bupivacaine in scalp block versus bupivacaine alone for postoperative pain management in patients undergoing craniotomy.

DETAILED DESCRIPTION:
Scalp block is proposed as a multimodal approach to preventing postoperative pain and hemodynamic responses to previous noxious stimulation during the operation.

The use of adjuvants, such as dexmedetomidine, a highly selective alpha-2 adrenergic receptor agonist, has recently been studied for its analgesic effects. Dexmedetomidine acts additionally to local anesthetics, prolonging their duration of action.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status I or II.
* Undergoing supratentorial elective planned craniotomies.

Exclusion Criteria:

* Patients refusal.
* History of known allergy to the used local anesthetic or dexmedetomidine.
* Bleeding disorders.
* Evidence of local infection at the site of injection.
* Emergency craniotomy.
* Psychotic disorder.
* Patients who will not be extubated in the operating room after surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative postoperative morphine consumption | 24 hours postoperatively
  If the Visual Analogue Scale (VAS) score is ≥3, rescue analgesia will be administered; intravenous morphine will be given at a dose of 0.05 mg/kg

SECONDARY OUTCOMES:
Mean arterial pressure | 24 hours postoperatively
  Mean arterial pressure will be measured at baseline, before Mayfield placement, 5 minutes after Mayfield insertion, at the end of surgery, and postoperatively at 2, 4, 6,12, and 24 hours postoperatively.
Heart rate | 24 hours postoperatively
  Heart rate will be measured at baseline, before Mayfield placement, 5 minutes after Mayfield insertion, at the end of surgery, and 2, 4, 6, 12, and 24 hours postoperatively.
Degree of pain | 24 hours postoperatively
  Pain intensity will be evaluated on a 0-10 visual analog scale (VAS). The VAS consists of a 10 cm line, with two endpoints representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). The VAS score will be recorded at baseline (after admission to PACU), then after 1 hour, 2 hours, 4 hours, 6 hours, 12 hours, and 24 hours postoperatively.
Time for 1st rescue analgesia | 24 hours postoperatively
  Time for 1st rescue analgesia will be recorded from the end of surgery till first dose of morphine administrated.
Incidence of complications | 24 hours postoperatively
  Incidence of complications such as postoperative nausea and vomiting, respiratory depression, or any other complication will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.